CLINICAL TRIAL: NCT01669785
Title: NUPRO Sensodyne Prophylaxis Paste With NovaMin for the Treatment of Dentin Hypersensitivity.
Brief Title: NUPRO Sensodyne Prophylaxis Paste With NovaMin Sensitivity Relief Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dentsply International (Industry)
Responsible Party: Sponsor
Organization: Dentsply Sirona Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTP-002
Record Dates: First submitted 2012-06-08; First posted 2012-08-21 (Estimated); Results first posted 2014-08-21 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Tooth Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group C (Active Comparator): NUPRO Classic Prophy Paste
  Administered on day one only. Unit dose cup contained enough paste for a single procedure. Contains no Novamin or Fluoride..
  Leave in contact for 60 seconds, rinse with water and expectorate.
  Interventions: Device: Group C
- Group A (Experimental): NUPRO Sensodyne Prophy Paste w/ Novamin
  Administered on day one only. Unit dose cup contained enough paste for a single procedure. Contains 15% Novamin. Does not contain Fluoride.
  Leave in contact for 60 seconds, rinse with water and expectorate
  Interventions: Device: Group B
- Group B (Experimental): NUPRO Sensodyne Prophy Paste w/ Novamin w/ Fluoride
  Administered on day one only. Unit dose cup contained enough paste for a single procedure. Contains 1.23% fluoride ion and 15% Novamin.
  Leave in contact for 60 seconds, rinse with water and expectorate.
  Interventions: Device: Group A

INTERVENTIONS:
Device: Group C — Abrasive, flavored dental prophylaxis paste for cleaning and polishing teeth.
  Other Names: NUPRO Classic Prophy Paste
  Arms: Group C
Device: Group A — Abrasive, flavored dental prophylaxis paste for cleaning and polishing teeth.
  Other Names: NUPRO Sensodyne Prophy Paste with NovaMin with Fluoride.
  Arms: Group B
Device: Group B — Abrasive, flavored dental prophylaxis paste for cleaning and polishing teeth.
  Other Names: NUPRO Sensodyne Prophy Paste with NovaMin without Fluoride.
  Arms: Group A

SUMMARY:
The study is intended to verify through clinical measurement that the NUPRO Sensodyne Prophylaxis Paste with Novamin provides immediate sensitivity relief as well as extended relief up to 28 days.

DETAILED DESCRIPTION:
It is hypothesized that the prophy paste with Novamin will give patients immediate sensitivity relief, as well as sensitivity relief up to 4 weeks (28 days) after measurement.

ELIGIBILITY:
Inclusion Criteria:

* Availability to complete in the 28 day duration.
* Two sensitive teeth, which are not adjacent to each other and preferably in different quadrants, which demonstrate cervical erosion, abrasion and gingival recession.
* Qualifying response to tactile stimuli as defined by a score of </= 20 grams.
* Qualifying response to air blast stimuli as defined by a score of >/= 1 on the Schiff Cold Air Sensitivity Scale.
* Subjects need to satisfy the qualifying response to stimuli for both parameters assesses (Tactile or Air Blast) on at least two teeth (non-adjacent) to be entered into the study.
* Good general health with no known allergies to products being tested.
* Use of a non-desensitizing dentifrice for 2 weeks prior to entry into the study.
* Subjects must have a minimum of 10 natural teeth, excluding 3rd molars.

Exclusion Criteria:

* Individuals who exhibit gross oral pathology.
* Females who may be pregnant or lactating or intending to become pregnant.
* Individuals who require anesthetic during scaling.
* Dental pathology which may cause pain similar to tooth sensitivity.
* Individuals with large amounts of calculus.
* Subjects with active infectious diseases such as hepatitis, HIV, or tuberculosis.
* Any condition requiring antibiotic prophylaxis for dental treatment.
* Excessive gingival inflammation.
* Individuals who had their teeth cleaned within 30 days of the screening appointment.
* Individuals who have had desensitizing treatment or tooth bleaching within 90 days of screening appointment.
* Oral pathology, chronic disease, or history of allergy to test products.
* Advanced periodontal disease or treatment for periodontal disease (including surgery) within the past twelve months.
* Sensitive teeth with mobility greater than one.
* Teeth with extensive/defective restorations (including prosthetic crowns), suspected pulpitis, caries, cracked enamel, or used as abutments for removable partial dentures.
* Regular use of sedatives, anti-inflammatory drugs, or analgesic.
* Participation in a desensitizing dentifrice study or regular use of a desensitizing dentifrice within the past 4 weeks.
* Current participation in any other clinical study or receipt of an investigational drug within 30 days of the screening visit at the start of the study.
* Personnel; a) an employee of the sponsor; b0 A member or relative of teh study site staff directly involved with the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2012-03; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Milleman, DDS, MPA, Principal Investigator — Salus Research
Locations (1):
- Salus Research, Inc., Fort Wayne, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A | Group B | Group C
Started | 45 | 48 | 46
Completed | 45 | 48 | 46
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group A: NUPRO Sensodyne Prophy Paste w/ Novamin. Administered on day one only.Unit dose cup contained enough paste for a single procedure. Contains 15% Novamin. Does not contain Fluoride.
  Leave in contact for 60 seconds, rinse with water and expectorate.
- Group B: NUPRO Sensodyne Prophy Paste w/ Novamin w/ Fluoride.Administered on day one only.Unit dose cup contained enough paste for a single procedure. Contains 1.23% fluoride ion and 15% Novamin.
  Leave in contact for 60 seconds, rinse with water and expectorate.
- Group C: NUPRO Classic Prophy Paste.Administered on day one only.Unit dose cup contained enough paste for a single procedure. Contains no Novamin or Fluoride.Leave in contact for 60 seconds, rinse with water and expectorate.
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Total
Number analyzed (Participants) | 45 | 48 | 46 | 139
Age, Customized [Mean (Standard Deviation); unit: mean years of age] | 44 (11.18274) | 41 (11.21829) | 43 (10.928) | 43 (11.10967)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 39 | 35 | 110
  Male | 9 | 9 | 11 | 29
Region of Enrollment [Number; unit: participants]
  United States | 45 | 48 | 46 | 139

OUTCOME MEASURES:

1. Primary Outcome: Baseline Pre-Prophy Assessment (Tactile Sensitivity)
Description: Pre-prophy procedure baseline assessment is measured with an electronic force sensing probe (Yeaple probe). Grams of force needed to elicit pain are recorded as hypersensitivity score for the tooth. 10,20,30,40, up to 50 grams of force are applied to the hypersensitive tooth until pain is elicited. The higher the score (the more grams of force needed to elicit a response of pain), the lower the hypersensitiv
  Subjects were required to have two sensitive teeth which are not adjacent to each other and preferably in different quadrants. Scores were obtained by taking the average over the scores for the evaluated teeth.
Time Frame: Pre-treatment measurement
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 45 | 48 | 46
grams | 10.56 (1.59) | 10.00 (0.00) | 10.98 (2.27)

2. Primary Outcome: Immediate Sensitivity Relief (Tactile Sensitivity)
Description: Assessment of sensitivity score via tactile and air blast measurements immediately after treatment. Tactile hypersensitivity is measured with an electronic force sensing probel (Yeaple probe). Grams of force needed to elicit pain are recorded as hypersensitivity score for the tooth. Grams of force needed to elicit pain are recorded as hypersensitivity score for the tooth. 10, 20, 30, 40 up to 50 grams of force are applied to the hypersensitive tooth until pain is elicited. The higher the score (the more grams of force needed to elicit a response of pain), the lower the hypersensitivity.
  Subjects were required to have two sensitive teeth which are not adjacent to each other and preferably in different quadrants. Scores were obtained by taking the average over the scores for the evaluated teeth.
Time Frame: Immediately after treatment .
Measure: Mean (Standard Deviation); unit: grams
Groups:
- Group A; Group B: NUPRO Sensodyne Prophy Paste w/ Novamin w/ Fluoride
  Administered on day one only. Unit dose cup contained enough paste for a single procedure. Contains 1.23% fluoride ion and 15% Novamin.
  Leave in contact for 60 seconds, rinse with water and expectorate.
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 45 | 48 | 46
grams | 19.61 (11.31) | 16.67 (9.01) | 12.01 (5.52)

3. Primary Outcome: Long-term Sensitivity Relief (Tactile Sensitivity)
Description: Assessment of sensitivity score via tactile measurements long term after treatment.
  Tactile hypersensitivity is measured with an electronic force sensing probel (Yeaple probe). Grams of force needed to elicit pain are recorded as hypersensitivity score for the tooth. Grams of force needed to elicit pain are recorded as hypersensitivity score for the tooth. 10 to 50 grams of force are applied to the hypersensitive tooth until pain is elicited. The higher the score (the more grams of force needed to elicit a response of pain), the lower the hypersensitivity.
  Subjects were required to have two sensitive teeth which are not adjacent to each other and preferably in different quadrants. Scores were obtained by taking the average over the scores for the evaluated teeth.
Time Frame: 28 days (+/- 2 days) post treatment.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 45 | 48 | 46
grams | 19.89 (11.46) | 16.51 (10.35) | 12.07 (5.20)

4. Secondary Outcome: Sensitivity Relief (Self-Assessment)
Description: All subjects completed a questionnaire titled "How sensitive are your teeth?" to assess their whole-mouth tooth sensitivity prior to the baseline assessments.
  The questionnaire contained a 4-item verbal descriptor scale as follows:
  Score 0= no discomfort or awareness of sensitivity; 1=mild discomfort/pain from sensitive teeth; 2=moderate discomfort/pain from sensitive teeth; 3=severe pain from sensitive teeth.
  The higher the score, the higher the hypersensitivity.
  Subjects were required to have two sensitive teeth which are not adjacent to each other and preferably in different quadrants. Scores were obtained by taking the average over the scores for the evaluated teeth.
Time Frame: Pre-Treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 45 | 48 | 46
units on a scale | 0.82 (0.72) | 0.67 (0.75) | 0.76 (0.74)

5. Primary Outcome: Baseline Pre-Prophy Assessment (Air Blast Sensitivity)
Description: Pre-prophy procedure baseline assessment using Schiff Cold Air Sensitivity scale (0-3).
  Air blast hypersensitivity is measured using the Schiff Cold Air Sensitivty scale (0-3). The scale is scored as follows:
  0=Subject does not respond to stimulus; 1= Subject responds to stimulus but does not request discontinuation of stimulus; 2=Subject responds to stimulus and requests discontinuation or moves from air stimulus; 3=Subject responds to stimulus, considers it painful and requests discontinuation.
  The higher the score, the higher the hypersensitivity.
  Subjects were required to have two sensitive teeth which are not adjacent to each other and preferably in different quadrants. Scores were obtained by taking the average over the scores for the evaluated teeth.
Time Frame: Pre-treatment measurement
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 45 | 48 | 46
units on a scale | 1.72 (0.58) | 1.70 (0.58) | 1.65 (0.60)

6. Primary Outcome: Immediate Sensitivity Relief (Schiff Air Blast Sensitivity)
Description: Assessment of sensitivity score via air blast measurements immediately after treatment.
  Air blast hypersensitivity is measured using the Schiff Cold Air Sensitivity scale (0-3). The scale is scored as follows:
  0=Subject does not respond to stimulus; 1= Subject responds to stimulus but does not request discontinuation of stimulus; 2=Subject responds to stimulus and requests discontinuation or moves from air stimulus; 3=Subject responds to stimulus, considers it painful and requests discontinuation.
  Subjects were required to have two sensitive teeth which are not adjacent to each other and preferably in different quadrants. Scores were obtained by taking the average over the scores for the evaluated teeth.
Time Frame: Immediately after treatment .
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 45 | 48 | 46
units on a scale | 0.88 (0.64) | 0.97 (0.52) | 1.72 (0.70)

7. Primary Outcome: Long-term Sensitivity Relief (Schiff Air Blast Sensitivity)
Description: Assessment of sensitivity score Schiff air blast measurements long term after treatment.
  Air blast hypersensitivity is measured using the Schiff Cold Air Sensitivity scale (0-3). The scale is scored as follows:
  0=Subject does not respond to stimulus; 1= Subject responds to stimulus but does not request discontinuation of stimulus; 2=Subject responds to stimulus and requests discontinuation or moves from air stimulus; 3=Subject responds to stimulus, considers it painful and requests discontinuation.
  Subjects were required to have two sensitive teeth which are not adjacent to each other and preferably in different quadrants. Scores were obtained by taking the average over the scores for the evaluated teeth.
Time Frame: 28 days (+/- 2 days) post treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 45 | 48 | 46
units on a scale | 0.87 (0.63) | 1.11 (0.61) | 1.67 (0.67)

8. Secondary Outcome: Post- Scaling Sensitivity Relief (Self-Assessment)
Description: All subjects completed a questionnaire titled "How sensitive are your teeth?" to assess their whole-mouth tooth sensitivity immediately following the scaling procedure.
  The questionnaire contained a 4-item verbal descriptor scale as follows:
  Score 0= no discomfort or awareness of sensitivity; 1=mild discomfort/pain from sensitive teeth; 2=moderate discomfort/pain from sensitive teeth; 3=severe pain from sensitive teeth.
  The higher the score, the higher the hypersensitivity.
  Subjects were required to have two sensitive teeth which are not adjacent to each other and preferably in different quadrants. Scores were obtained by taking the average over the scores for the evaluated teeth.
Time Frame: Post-scaling procedure,immediate
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 45 | 48 | 46
units on a scale | 1.31 (0.79) | 0.98 (0.67) | 1.28 (0.72)

9. Secondary Outcome: Post-prophylaxis Sensitivity Relief (Self-Assessment)
Description: All subjects completed a questionnaire titled "How sensitive are your teeth?" to assess their whole-mouth tooth sensitivity immediately following the timed, 1-minute prophylaxis paste application.
  The questionnaire contained a 4-item verbal descriptor scale as follows:
  Score 0= no discomfort or awareness of sensitivity; 1=mild discomfort/pain from sensitive teeth;2=moderate discomfort/pain from sensitive teeth; 3=severe pain from sensitive teeth.
  The higher the score, the higher the hypersensitivity.
  Subjects were required to have two sensitive teeth which are not adjacent to each other and preferably in different quadrants. Scores were obtained by taking the average over the scores for the evaluated teeth.
Time Frame: Immediately following post-prophylaxis treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 45 | 48 | 46
units on a scale | 1.00 (0.90) | 0.90 (0.81) | 1.09 (0.69)

10. Secondary Outcome: Long-term Sensitivity Relief (Self-Assessment)
Description: All subjects completed a questionnaire titled "How sensitive are your teeth?" to assess their whole-mouth tooth sensitivity 28 days following prophylaxis treatment.
  The questionnaire contained a 4-item verbal descriptor scale as follows:
  Score 0= no discomfort or awareness of sensitivity;1=mild discomfort/pain from sensitive teeth; 2=moderate discomfort/pain from sensitive teeth; 3=severe pain from sensitive teeth.
  The higher the score, the higher the hypersensitivity.
  Subjects were required to have two sensitive teeth which are not adjacent to each other and preferably in different quadrants. Scores were obtained by taking the average over the scores for the evaluated teeth.
Time Frame: 28 days post-prophylaxis treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 45 | 48 | 46
units on a scale | 0.60 (0.62) | 0.50 (0.71) | 0.72 (0.69)

ADVERSE EVENTS:
Time Frame: Patients were monitored for adverse events during intraoral examinations performed after paste application and 28 days following paste application.
Arm/Group | Group A | Group B | Group C
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/48 | 0/46
Other Adverse Events (participants affected / at risk) | 0/45 | 0/48 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less